CLINICAL TRIAL: NCT00567515
Title: Safety and Effectiveness of Left Atrial Appendage Occlusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUS 2007-1
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LAA Clip (Experimental): AtriCure LAA Exclusion System
  Interventions: Device: AtriCure LAA Exclusion System

INTERVENTIONS:
Device: AtriCure LAA Exclusion System — Placement of clip of LAA.

SUMMARY:
This study is to evaluate acute and long-term safety and effectiveness of Left atrial appendage occlusion (LAA)with the AtriCure LAA Occlusion System. This device will be applied in patients with atrial fibrillation (AF), paroxysmal, persistent and permanent, undergoing cardiac surgery with a concomitant Maze/Ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Documented history (paroxysmal, persistent or permanent) of AF [one episode within the last 12 months of enrollment]
2. Elective Maze procedure
3. Suitable anatomy
4. Able and willing to sign informed consent
5. Age over 18 years

Exclusion Criteria:

1. Patient from Intensive Care Unit with either:

   1. intra-venous catecholamines
   2. ventilator
   3. cardiac index <1.8 l/min.
2. Reoperative Cardiac Surgery
3. Systemic or Inflammatory disease
4. Dialysis
5. Recent myocardial infarction (< 21 days)
6. History of pericarditis
7. Patient taking part in any other device or drug study
8. Patient with known sensitivity or allergy to any of the device components
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety - Device related complications | 30 days
Efficacy - Occlusion of the LAA | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Genoni, MD, Professor, Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Caliskan E, Sahin A, Yilmaz M, Seifert B, Hinzpeter R, Alkadhi H, Cox JL, Holubec T, Reser D, Falk V, Grunenfelder J, Genoni M, Maisano F, Salzberg SP, Emmert MY. Epicardial left atrial appendage AtriClip occlusion reduces the incidence of stroke in patients with atrial fibrillation undergoing cardiac surgery. Europace. 2018 Jul 1;20(7):e105-e114. doi: 10.1093/europace/eux211. PMID 29016813
- [Derived] Emmert MY, Puippe G, Baumuller S, Alkadhi H, Landmesser U, Plass A, Bettex D, Scherman J, Grunenfelder J, Genoni M, Falk V, Salzberg SP. Safe, effective and durable epicardial left atrial appendage clip occlusion in patients with atrial fibrillation undergoing cardiac surgery: first long-term results from a prospective device trial. Eur J Cardiothorac Surg. 2014 Jan;45(1):126-31. doi: 10.1093/ejcts/ezt204. Epub 2013 May 8. PMID 23657550
- [Derived] Salzberg SP, Plass A, Emmert MY, Desbiolles L, Alkadhi H, Grunenfelder J, Genoni M. Left atrial appendage clip occlusion: early clinical results. J Thorac Cardiovasc Surg. 2010 May;139(5):1269-74. doi: 10.1016/j.jtcvs.2009.06.033. Epub 2009 Nov 1. PMID 19880144